CLINICAL TRIAL: NCT01775280
Title: Radiologic, Histologic and Immunologic Response to Radioembolization of Hepatic Tumors
Brief Title: Response of Hepatic Tumors to Radioembolization
Acronym: RESRAD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USZ-ZH-VIS-RESRAD
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Hepatocellular Carcinoma; Intrahepatic Cholangiocarcinoma; Liver Metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radioembolization (Experimental): Radioembolization using Yttrium-90 microspheres using a transarterial approach
  Interventions: Radiation: Injection of Ytttrium-90 microspheres into the hepatic artery

INTERVENTIONS:
Radiation: Injection of Ytttrium-90 microspheres into the hepatic artery — INjection of Y-90 particles into the hepatic artery using endovascular access

SUMMARY:
The study enrolls patients with non-resectable or borderline resectable hepatocellular carcinoma (HCC), intraheaptic choalngiocarcinoma (IHCC) or colorectal cancer metastasis. Patients are not a candidates for liver transplantation and have only limited extrahepatic disease. All patients are treated with radioembolization. Primary endpoint is the percentage of patients that can be downstaged to resectability.

Secondary endpoints are radiologic response to radioembolization,tissue response to radiomembolization and systemic immune response and intra-tumoral T-cell response to radioembolization.

* Trial with radiotherapy

ELIGIBILITY:
Inclusion criteria: - Patients already considered for radioembolization fulfil criteria to be included in the study. If radioembolization is not considered by the tumor board, inclusion in the study should not be considered.

- Non-resectable or borderline resectable liver tumors (HCC, CRCM or CCC) as as-sessed by a multidisciplinary tumor-board. Non-resectability or borderline resectablily is based closeness to essential nonresectable structures (f.e. the portal vein bifurca- tion or hepatic vein trifurcation) or insufficient liver volume after resection, general performance status of the patient.

Chemotherapy (mostly applicable to CRCM) should be termininated at least 4 weeks prior to enrolling patients in the study.

* Concomitant manoevers to manipulate liver volume like portal vein embolization or ligation and two-stage resections are allowed
* Male or female patients 18-99 years of age
* Presentation of the case at the Multidisciplinary Meeting attended by hepatobiliary surgeons, oncologists, hepatologists and radiologists
* Written informed consent given by the patient
* Adequate liver function or kidney function tests, including any of the following. It is possible to perform endoscopic or percutaneous stent placement to achieve normal-isation of laboratory parameters.
* Women who are not breastfeeding and are using effective contraception if sexually active, who are not pregnant and agree not to become pregnant during the 12 months thereaf-ter. A negative pregnancy test before inclusion into the trial is required for women < 50 years. Men who agree not to father a child during participation in the trial or during the 12 months thereafter.
* Effective contraception

Patient compliance and geographic proximity

Exclusion criteria: -Patients with no clinical indications for radioembolization (resectable tumors, no need for downsizing)

* contraindications on ethical grounds,
* women who are pregnant or breast feeding,
* significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardi-ovascular disease, etc) as based on above mentioned labaratory values or preopera-tive cardiac assessment making the patient unsuitable for major surgery known or suspected non-compliance, drug or alcohol abuse, enrolment into a clinical trial within last 4 weeks, extrahepatic tumor burden, as evaluated by PET/CT or chest CT. Potentially resectable small lung nodules or hilar lymphadenopathy by CT or PET in case of MCRC mandate systemic chemotherapy prior to enrolment into this trial if not already performed. The patient may be en-rolled into this trial to be downstaged by radioembolization after finishing systemic chemotherapy.
* Anatomic variant in arteriogram which prevents selective delivery of the chemother-apy to the liver (discussed within group of principal investigators)
* Life expectancy < 3 months
* Candidacy for liver transplantation in the case of HCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint ist the percentage of patients that can be downstaged to resectability | 2012 to 2015

SECONDARY OUTCOMES:
Histologic response to radioembolization | 2012 to 2015
  Resected specimen will be examined for changes related to radioembolization like endothelial damage, necrosis, fibrosis
Immunological response to radioembolization | 2012 to 2015
  Circulating T-cells and tissue based T-cells will be examined for their response to tumor antigens, clonal proliferation.
  Serologic response to tumor antigens will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Erik Schadde, MD, Principal Investigator — University Hospital Zurich, Division of Visceral and Transplant Surgery; Niklaus Schaefer, MD, Principal Investigator — University Hospital Zurich, Division of Nuclear Medicine
Locations (1):
- University Hospital Zurich, Divisions of Visceral Surgery and Nucelar Medicine, Zurich, Canton of Zurich, Switzerland